CLINICAL TRIAL: NCT05501678
Title: Randomized Placebo-controlled Crossover Trial of Diphenhydramine for Sleep in Children With Autism
Brief Title: Trial of Diphenhydramine for Sleep in Children With Autism
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Antonio Hardan, Professor of Psychiatry and Behavioral Sciences, Stanford University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: IRB-66941; 1P50HD109861 (NIH)
Record Dates: First submitted 2022-08-12; First posted 2022-08-15 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Autism; Autism Spectrum Disorder
Keywords: Diphenhdramine; Sleep; clinical trial; autism
MeSH Terms: conditions — Autistic Disorder; Autism Spectrum Disorder | interventions — Diphenhydramine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Diphenhydramine, then Placebo (Experimental): Participants will first receive Diphenhydramine for a 4-week period. A 25 mg dose of Diphenhydramine will be given at bedtime for one week and then will increase to 50 mg if needed and if well tolerated.
  Participants will then receive Placebo (fake tablet) for a 4-week period. A 25 mg dose of matching Placebo will be given at bedtime for one week and then will increase to 50 mg if needed and if well tolerated.
  Interventions: Drug: Diphenhydramine; Drug: Placebo
- Placebo, then Diphenhydramine (Experimental): Participants will first receive Placebo (fake tablet) for a 4-week period. A 25 mg dose of matching Placebo will be given at bedtime for one week and then will increase to 50 mg if needed and if well tolerated.
  Participants will then receive Diphenhydramine for a 4-week period. A 25 mg dose of Diphenhydramine will be given at bedtime for one week and then will increase to 50 mg if needed and if well tolerated.
  Interventions: Drug: Diphenhydramine; Drug: Placebo

INTERVENTIONS:
Drug: Diphenhydramine — 25mg (and up to 50mg) Diphenhydramine given orally
  Other Names: Benadryl
Drug: Placebo — Matching Placebo given orally

SUMMARY:
The purpose of this study is to examine the effect of diphenhydramine on sleep in children and adolescents with Autism Spectrum Disorder (ASD). Diphenhydramine is an anti-histaminergic agent with strong hypnotic properties. To accomplish this, the investigators will use a randomized double-blind placebo-controlled crossover 8-week study design to examine the effect of diphenhydramine on sleep physiology as assessed by polysomnography (PSG), actigraphy, circadian rhythm, and clinical measures.

ELIGIBILITY:
Inclusion criteria:

Participants will meet the following

* Outpatients between 8 and 17 years of age at the time of consent
* Diagnostic and Statistical Manual, 5th edition (DSM-5) criteria for Autism Spectrum Disorder (ASD) on the basis of clinical evaluation, confirmed with the Autism Diagnostic Interview-Revised (ADI-R) and the Autism Diagnostic Observation Schedule, 2nd Ed (ADOS-2)
* Males and females
* Availability of polysomnography (PSG) or actigraphy data
* Sleep disturbances as assessed using Children's Sleep Habits Questionnaire (CSHQ) with a score of 41 or higher
* care provider who can reliably bring participant to clinic visits, provide trustworthy ratings, and interacts with participant on a regular basis
* stable medications for at least 2 weeks, with the exception of Prozac which is required to be stable for at least 4 weeks
* no planned changes in psychosocial and biomedical interventions during the trial
* willingness to provide additional saliva samples and participate in key study procedures (i.e., safety measurements every visit, PSG at weeks 4 and 8, and wear the actigraphy watch for 2 weeks before the beginning of trial as well as during the 8 weeks of the trial).

Exclusion criteria:

Participants will be excluded if one or more of the following is met

* active suicidal ideation or DSM-5 diagnosis of schizophrenia, schizoaffective disorder, or psychotic disorder
* active medical problems: migraine, asthma, seizure disorder, significant physical illness (e.g., anaphylaxis, serious liver, renal, or cardiac pathology)
* evidence of a metabolic, or infectious etiology for the participant's autism on the basis of medical history, neurologic history, and available tests for inborn errors of metabolism and chromosomal analysis
* pregnant or sexually active females not using a reliable method of contraception (urinary tests for pregnancy will be employed in this study)
* individuals taking benzodiazepines, antiepileptic medications when prescribed for seizure disorder/epilepsy, melatonin, and antihistamines
* history of hypersensitivity to diphenhydramine
* history of severe side effects from diphenhydramine
* history of adequate trial of diphenhydramine
* current use of any medications known to interact with diphenhydramine such as medications inhibiting CYP2D6
* taking anticholinergic agents (e.g., trihexyphenidyl, thioridazine).

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 26 (Estimated)
Dates: Start 2023-08-09 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in sleep latency as measured by polysomnography (PSG) and actigraphy | Baseline, Week 4 and Week 8
Change from baseline in duration of non-rapid eye movement (NREM) sleep as measured by polysomnography (PSG) | Baseline, Week 4 and Week 8

SECONDARY OUTCOMES:
Change from baseline in sleep efficiency as measured by polysomnography (PSG) and actigraphy | Baseline, Week 4 and Week 8

OTHER OUTCOMES:
Change from baseline on Children's Sleep Habits Questionnaire (CSHQ) subscale scores | Baseline, Week 4, Week 8
Change from baseline on Aberrant Behavior Checklist, Second Edition (ABC-2) subscale scores | Baseline, Week 4, Week 8
Change from baseline on Parent Sleep Habits Questionnaire Parent (PSHQ) scores | Baseline, Week 4, Week 8
Change from baseline on Clinical Global Impression Scale (CGI) scores | Baseline, Week 1, Week 2, Week 3, Week 4, Week 5, Week 6, Week 7, and Week 8
Change from baseline on Child Behavior Checklist (CBCL) scores | Baseline, Week 4, Week 8
Change from baseline on Social Responsiveness Scale, Second Edition (SRS-2) scores | Baseline, Week 4, Week 8
Change from baseline on Repetitive Behavior Scale - Revised (RBS-R) scores | Baseline, Week 4, Week 8
Change from baseline on Sensory Profile Questionnaire (SPQ) scores | Baseline, Week 4, Week 8
Change from baseline on Stanford Social Dimension Scale (SSDS) scores | Baseline, Week 4, Week 8
Change from baseline on Dimensional Assessment of Repetitive Behaviors (DARB) scores | Baseline, Week 4, Week 8
Change from baseline on NEuroPSYchological Assessment, 2nd Edition (NEPSY-2) Affect Recognition scores | Baseline, Week 4, Week 8

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Y. Hardan, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: Yes
We will submit de-identified clinical data to the NIMH Data Archive (NDA) data repository.
URL: https://nda.nih.gov/nda/data-contribution.html